CLINICAL TRIAL: NCT04709510
Title: Outcomes of Short-term Perioperative Thromboprophylaxis After Gastrointestinal Cancer Surgery
Brief Title: Short-term Perioperative Thromboprophylaxis After Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nuray COLAPKULU, Surgical Resident (Research Assistant) at General Surgery, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RetroThrombo
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; short-term thromboprophylaxis
MeSH Terms: conditions — Venous Thrombosis | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Intervention Model Description: Retrospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AllPatients (Other): There is only one cohort in this study. They all received the same follow up and ultrasound protocol.
  Interventions: Diagnostic Test: Duplex Ultrasound

INTERVENTIONS:
Diagnostic Test: Duplex Ultrasound — Duplex Ultrasound was performed for every participants for the diagnosis of symptomatic or asymptomatic deep vein thrombosis

SUMMARY:
Major abdominal surgery for cancer is major risk factor for thromboembolism. Patients who undergo major abdominal surgery are prone to develop venous thromboembolism, both in the early postoperative period and after hospital discharger. There are strong recommendations in the international guidelines in favor to pharmacological thromboprophylaxis. Thus there is no consensus dor the duration of the prophylaxis. There are authors that suggest extended prophylaxis up to 4 week after surgery. On the other hand, there are prospective randomized trials that inpatient (short-term up to 7-10 days) prophylaxis is adequate.

DETAILED DESCRIPTION:
This is a retrospective cohort study with 89 patients who underwent major abdominal surgery for colorectal and gastric cancer. All patients received short term prophylaxis (during hospital stay only) rather than extended prophylaxis (4 weeks). All participants received duplex ultrasound in the study period for the diagnosis of deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Major abdominal surgery gor colorectal or gastric cancer
* Caprini Risk score less than 9
* No history of anticoagulant treatment
* Thromboprophylaxis during hospital stay only

Exclusion Criteria:

* Younger than 18
* Caprini Risk score 9 and above
* History of anticogulants
* Not reachable by phone etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The incidence of thromboembolic events by radiological assessment | 3 years follow up
  All patients in the cohort received short time prophylaxis for deep vein thrombosis instead of prolonged duration. All patients will be assessed with ultrasound.

SECONDARY OUTCOMES:
Rate of predisposing factors of the patients | 3 years follow up
  The patients with deep vein thrombosis in the cohort will be assessed according to their postoperative period features, histories, chemo treatments etc. with and questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Alimoglu, Prof, Study Chair — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No